CLINICAL TRIAL: NCT03276052
Title: A Phase I, Open-Label, Single and Multiple Dose (Twice-Daily), Clinical Trial to Evaluate the Pharmacokinetics, Safety and Tolerability of Aclidinium Bromide 400 μg Administered by Inhalation in Healthy Chinese Participants
Brief Title: A Phase I, Open-Label, Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Aclidinium Bromide in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6572C00002; M-AS273-01 (Other: Clinical Trial Protocol Code)
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics
MeSH Terms: interventions — aclidinium bromide

STUDY DESIGN:
Intervention Model Description: Single and Multiple Dose (Twice-Daily)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aclidinium Bromide 400 μg (Experimental): One inhalation from the 400 μg Aclidinium Bromide inhaler.
  Interventions: Drug: Aclidinium Bromide 400 μg

INTERVENTIONS:
Drug: Aclidinium Bromide 400 μg — Aclidinium Bromide 400 μg BID inhalation powder. One oral inhalation via Genuair® dry powder inhaler (DPI)

SUMMARY:
A Phase I, single centre, open-label study to investigate the pharmacokinetics (PK), safety and tolerability of single and multiple twice daily doses of inhaled Aclidinium Bromide in healthy Chinese male and female subjects.

DETAILED DESCRIPTION:
Screening will be performed within 21 days of dosing on Day 1. Eligible participants will be admitted to the trial center on Day -1.

Subjects will receive single dose on Day 1, twice daily regimen is from D5 to D8, and only morning dose will be given on Day 9.

During treatment period, from Day 1 through Day 11 at Visit 2, safety measurements (blood pressure, 12-lead ECG; and AE/SAE monitoring) and blood samples for PK assessments will be collected at predetermined time points.

Clinical laboratory tests (haematology, serum biochemistry and urinalysis) will be performed under fasting conditions at Day -1 at Visit 2.

A follow-up visit will be performed on Day 15.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to communicate with medical team and staff, willing to participate in the trial, willing to give written informed consent, and comply with the trial restrictions.
2. Healthy subjects: Chinese men or non-pregnant, non-lactating women, 18 through 45 years old at Visit 1 (Screening).
3. Have a body mass index (BMI) ≥19 kg/m2 and ≤ 26 kg/m2
4. Resting heart rate ≥ 50 beats per minute (bpm) and ≤ 100 bpm at Visit 1 (Screening) and at admission to the unit on Day -1 at Visit 2.
5. Non-smoker (never smoked or has not smoked within 2 years prior to the first dose of investigational product [IP]).
6. Demonstrate satisfactory technique in the use of the DPI at screening.

Exclusion Criteria:

1. History of any significant drug allergy or hypersensitivity to aclidinium bromide or other muscarinic antagonists.
2. Have abnormal and clinically significant results on the physical examination, medical history, serum biochemistry, haematology, or urinalysis at Visit 1 (Screening).
3. Sustained resting systolic blood pressure ≥ 140 or ≤ 90 mmHg and resting diastolic blood pressure ≥ 90 or ≤ 50 mmHg at Visit 1 (Screening) or Day -1 at Visit 2.
4. Electrocardiogram (ECG) showing corrected QT interval (QTc) using Fridericia's correction (QTcF) ≥ 450 msec for male participants and ≥460 msec for female participants as indicated in the centralised reading report assessed at Screening (Visit 1).
5. Have a history of alcohol or substance abuse within the previous 5 years, as reported by the participants.
6. Positive results for drugs of abuse at Visit 1 (Screening).
7. Positive test for hepatitis B surface antigen (HBsAg), hepatitis C antibody and/or human immunodeficiency virus (HIV) antibodies at Visit 1 (Screening).
8. Use of any medication within 2 weeks or within the equivalent time of 5 half-lives of taking the last dose (whichever is longer) before the first dose of IP, or hormonal drug products and traditional Chinese medicines within 30 days before the first dose of IP.
9. Have consumed caffeine or any grapefruit-containing products within 48 hours or alcohol within 72 hours before Day -1.
10. Participation in any other clinical investigation using an experimental drug requiring repeated blood or plasma draws within 60 days of Day 1 at Visit 2.
11. Have participated in a blood/plasma donation or blood loss greater than 400 mL within 90 days, or greater than 200 mL within 30 days prior to screening (Visit 1).
12. Recent history of a disease or condition that would result in any residual upper respiratory airways/lung inflammatory process or residual limited lung function at the time of Day 1 at Visit 2.
13. History of confirmed COVID-19 infection.
14. Have any gastrointestinal, hepatic, or renal condition that might affect the absorption, distribution, biotransformation, or excretion of aclidinium bromide.
15. Inability to be venipunctured or tolerate venous access as determined by the PI or designee.
16. Participants unable to give their consent, or participants of consenting age but under guardianship, or vulnerable participants.
17. In the opinion of the PI, participants who are unlikely to comply with the protocol requirements, instructions, and trial-related restrictions.
18. Participant is a relative of the Investigator or any sub-investigator, research assistant, pharmacist, trial coordinator, or other staff or directly involved in the conduct of the clinical trial.
19. Any other conditions that, in the Investigator's opinion, might have indicated the participant to be unsuitable for the study (e.g. confirmed/suspected COVID-19)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Li, Principal Investigator — West China Hostial, Sichuan University
Locations (1):
- Research Site, Chengdu, China

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6572C00002&attachmentIdentifier=34bbcc6d-dc20-44c5-b0de-95fd4447d5f1&fileName=D6572C00002_CSR_Synopsis_Final_Client_Redacted.pdf&versionIdentifier=
- See also: Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6572C00002&attachmentIdentifier=8883e55e-3d16-4b5a-b238-3d14d7889d5e&fileName=D6572C00002_Protocol_Final_Client_Redacted.pdf&versionIdentifier=
- See also: Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6572C00002&attachmentIdentifier=0de469e8-b9f2-421f-825b-a376882879f5&fileName=D6572C00002_Statistical_analysis_plan_Final_Client_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at one study centre in China between 14 October 2021 to 26 November 2021.
Pre-assignment Details: The Screening period was of 21 days before randomization. Participants who met the inclusion and none of the exclusion criteria were enrolled to the study. All study assessments were performed as per the schedule of assessment.
Groups:
- Aclidinium Bromide 400 μg: Healthy Chinese participants received aclidinium bromide 400 μg.
Period: Overall Study
Arm/Group | Aclidinium Bromide 400 μg
Started | 43
Completed | 20
Not Completed | 23
Not completed — Withdrawal by Subject | 5
Not completed — Screening failure (non-fulfilment of inclusion/exclusion criteria) | 18

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of IP and for whom any safety post-dose data were available.
Arm/Group | Aclidinium Bromide 400 μg
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.15 (5.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Chinese | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Characterization of Cmax, taken directly from the individual concentration-time curve after single dose or multiple dose.
Time Frame: Day 1 and Day 9
Population: The PK analysis set consisted of all participants in the safety analysis set who received at least 1 dose of aclidinium bromide.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- Single Dose (Day 1): Healthy Chinese participants received a single dose of aclidinium bromide 400 μg on Day 1.
- Multiple Dose (Day 9): Healthy Chinese participants received twice daily doses of aclidinium bromide from Day 5 to Day 8, followed by a single dose on Day 9.
Arm/Group | Single Dose (Day 1) | Multiple Dose (Day 9)
Number analyzed (Participants) | 20 | 20
pg/mL
  Aclidinium bromide | 238.6 (51.67) | 341.3 (40.24)
  LAS34850 (inactive acid metabolite) | 3831 (24.99) | 4891 (16.52)
  LAS34823 (inactive alcohol metabolite) | 164.0 (45.05) | 294.1 (39.93)

2. Primary Outcome: Time to Reach Maximum Observed Concentration (Tmax)
Description: Characterization of Tmax, taken directly from the individual concentration-time curve after single dose or multiple dose.
Time Frame: Day 1 and Day 9
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Single Dose (Day 1) | Multiple Dose (Day 9)
Number analyzed (Participants) | 20 | 20
Hour
  Aclidinium bromide | 0.08 [0.08 to 0.10] | 0.08 [0.08 to 0.10]
  LAS34850 (inactive acid metabolite) | 3.00 [2.00 to 3.00] | 2.50 [1.50 to 3.00]
  LAS34823 (inactive alcohol metabolite) | 0.08 [0.08 to 0.50] | 0.08 [0.08 to 0.50]

3. Primary Outcome: Area Under the Concentration-time From Zero to Infinity (AUCinf)
Description: Characterization of AUCinf (single dose). Area under the concentration time curve from time zero extrapolated to infinity. AUC(0-∞) is estimated by AUC(last) + Clast/λz where Clast is the last observed quantifiable concentration.
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Single Dose (Day 1)
Number analyzed (Participants) | 20
h*pg/mL
  Aclidinium bromide | 266.1 (59.15)
  LAS34850 (inactive acid metabolite) | 29970 (17.63)
  LAS34823 (inactive alcohol metabolite) | 684.4 (48.04)

4. Primary Outcome: Area Under the Concentration-time From Time 0 to 12 Hours Post-dose [AUC(0-12)]
Description: The AUC(0-12) of aclidinium bromide and its metabolites after single dose of aclidinium bromide in healthy Chinese participants is investigated. Description of the AUC(0-12), partial area under the concentration- time curve in the dose interval after single dose or multiple dose.
Time Frame: Day 1 and Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Single Dose (Day 1) | Multiple Dose (Day 9)
Number analyzed (Participants) | 20 | 20
h*pg/mL
  Aclidinium bromide | 167.1 (40.19) | 357.8 (32.28)
  LAS34850 (inactive acid metabolite) | 22730 (18.64) | 33910 (15.33)
  LAS34823 (inactive alcohol metabolite) | 438.1 (37.26) | 1031 (25.56)

5. Primary Outcome: Area Under the Concentration-time From Zero to the Last Quantifiable Concentration (AUClast)
Description: Characterization of AUClast, taken directly from the individual concentration-time curve after single dose or multiple dose.
Time Frame: Day 1 and Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Single Dose (Day 1) | Multiple Dose (Day 9)
Number analyzed (Participants) | 20 | 20
h*pg/mL
  Aclidinium bromide | 208.9 (57.23) | 609.4 (36.49)
  LAS34850 (inactive acid metabolite) | 29010 (18.02) | 50370 (16.78)
  LAS34823 (inactive alcohol metabolite) | 550.4 (54.05) | 1849 (25.49)

6. Primary Outcome: Half-life Associated With Terminal Slope of a Semi-logarithmic Concentration-time Curve (t½λz)
Description: Characterization of t½λz, of aclidinium bromide and its metabolites after single and multiple doses of aclidinium bromide in healthy Chinese participants.
Time Frame: Day 1 and Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Single Dose (Day 1) | Multiple Dose (Day 9)
Number analyzed (Participants) | 20 | 20
Hour
  Aclidinium bromide | 13.50 (91.55) | 21.42 (25.63)
  LAS34850 (inactive acid metabolite) | 8.322 (26.83) | 12.68 (18.98)
  LAS34823 (inactive alcohol metabolite) | 9.964 (42.98) | 17.66 (12.35)

7. Primary Outcome: Apparent Total Body Clearance From Plasma After Extravascular Administration (CL/F)
Description: Characterization of CL/F, of aclidinium bromide after single and multiple doses of aclidinium bromide in healthy Chinese participants.
Time Frame: Day 1 and Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Single Dose (Day 1) | Multiple Dose (Day 9)
Number analyzed (Participants) | 20 | 20
Liter/hour | 1503 (59.15) | 1118 (32.28)

8. Primary Outcome: Volume of Distribution (Apparent) Following Extravascular Administration Based on Terminal Phase (Vz/F)
Description: Characterization of Vz/F, of aclidinium bromide after single and multiple doses of aclidinium bromide in healthy Chinese participants.
Time Frame: Day 1 and Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Single Dose (Day 1) | Multiple Dose (Day 9)
Number analyzed (Participants) | 20 | 20
Liter | 29280 (45.53) | 34550 (40.89)

9. Primary Outcome: Mean Residence Time of the Unchanged Drug in the Systemic Circulation (MRTinf)
Description: Characterization of MRTinf, of aclidinium bromide after single dose of aclidinium bromide in healthy Chinese participants.
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Single Dose (Day 1)
Number analyzed (Participants) | 20
Hour | 13.45 (95.18)

10. Primary Outcome: Minimum Observed Drug Concentration (Cmin)
Description: Characterization of Cmin, taken directly from the individual concentration-time curve after single dose or multiple dose.
Time Frame: Day 1 and Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Single Dose (Day 1) | Multiple Dose (Day 9)
Number analyzed (Participants) | 20 | 20
pg/mL
  Aclidinium bromide | 3.251 (56.25) | 11.55 (41.22)
  LAS34850 (inactive acid metabolite) | 647.8 (20.84) | 1223 (19.34)
  LAS34823 (inactive alcohol metabolite) | 14.82 (31.53) | 43.03 (28.55)

11. Primary Outcome: Average Drug Concentration Over a Dosing Interval (Cavg)
Description: Characterization of Cavg, of aclidinium bromide and its metabolites after multiple doses of aclidinium bromide in healthy Chinese participants.
Time Frame: Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Multiple Dose (Day 9)
Number analyzed (Participants) | 20
pg/mL
  Aclidinium bromide | 29.82 (32.28)
  LAS34850 (inactive acid metabolite) | 2826 (15.33)
  LAS34823 (inactive alcohol metabolite) | 85.95 (25.56)

12. Primary Outcome: Accumulation Ratio for Cmax [Rac(Cmax)]
Description: Characterization of Rac(Cmax), of aclidinium bromide and its metabolites after multiple doses of aclidinium bromide in healthy Chinese participants. Rac(Cmax) is caculated as a ratio for Cmax estimated as (ratio of Css,max on Day 9/Cmax on Day 1).
Time Frame: Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Groups:
- Aclidinium Bromide 400 μg: Healthy Chinese participants received twice daily doses of aclidinium bromide from Day 5 to Day 8, followed by a single dose on Day 9.
Arm/Group | Aclidinium Bromide 400 μg
Number analyzed (Participants) | 20
Ratio
  Aclidinium bromide | 1.431 (44.18)
  LAS34850 (inactive acid metabolite) | 1.277 (20.40)
  LAS34823 (inactive alcohol metabolite) | 1.794 (45.61)

13. Primary Outcome: Accumulation Ratio for Cmin (Rac[Cmin])
Description: Characterization of Rac(Cmin), of aclidinium bromide and its metabolites after multiple doses of aclidinium bromide in healthy Chinese participants. Rac(Cmin) is calculated as ratio for Cmin estimated as (ratio of Css, Cmin on Day 9/ Cmin on Day 1)
Time Frame: Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Aclidinium Bromide 400 μg
Number analyzed (Participants) | 20
Ratio
  Aclidinium bromide | 3.554 (50.32)
  LAS34850 (inactive acid metabolite) | 1.888 (22.90)
  LAS34823 (inactive alcohol metabolite) | 2.903 (37.70)

14. Primary Outcome: Accumulation Ratio for AUCτ (Rac[AUC])
Description: Characterization of Rac(AUC), of aclidinium bromide and its metabolites after multiple doses of aclidinium bromide in healthy Chinese participants. Rac(AUC), calculated as ratio of AUC(0-12) on day 9 and AUC0-12 on Day 1.
Time Frame: Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Aclidinium Bromide 400 μg
Number analyzed (Participants) | 20
Ratio
  Aclidinium bromide | 2.141 (37.64)
  LAS34850 (inactive acid metabolite) | 1.492 (16.84)
  LAS34823 (inactive alcohol metabolite) | 2.354 (40.94)

15. Primary Outcome: Fluctuation Index During a Dosing Interval (%Fluc)
Description: Characterization of %Fluc, of aclidinium bromide and its metabolites after multiple doses of aclidinium bromide in healthy Chinese participants. The %Fluc index is estimated as 100 x (Cmax- Cmin)/Cav.
Time Frame: Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Multiple Dose (Day 9)
Number analyzed (Participants) | 20
Percentage
  Aclidinium bromide | 1102 (34.70)
  LAS34850 (inactive acid metabolite) | 128.9 (14.90)
  LAS34823 (inactive alcohol metabolite) | 289.2 (35.31)

16. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The safety, and tolerability of aclidinium bromide 400 μg BID after single and multiple dose administration in healthy Chinese participants was evaluated.
Time Frame: From Screening (Day -21 to Day -2) until the follow-up visit (Day 15)
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Aclidinium Bromide 400 μg
Number analyzed (Participants) | 20
Participants
  Any AE | 5
  Any AE with outcome = death | 0
  Any SAE (including events with outcome = death) | 0
  Any AE leading to discontinuation of IP | 0
  Any AE of special interest | 1

ADVERSE EVENTS:
Time Frame: From Screening (Day -21 to Day -2) until the follow-up visit (Day 15)
Arm/Group | Aclidinium Bromide 400 μg
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aclidinium Bromide 400 μg (N=20)
Syncope (Nervous system disorders) | 1 (1)
Atrial escape rhythm (Cardiac disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT03276052/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT03276052/SAP_001.pdf